CLINICAL TRIAL: NCT06838286
Title: A Multicenter, Prospective, Non-interventional Observation Study to Evaluate the Safety and Effectiveness of OAD Triple Therapy in Korean Type 2 Diabetic Mellitus Patients
Brief Title: Korean Study on Safety and Effectiveness of OAD Triple Therapy in Type 2 Diabetes
Acronym: TRIO
Status: Recruiting | Type: Observational
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: D141_01DM2303
Record Dates: First submitted 2024-06-30; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Korean patients; Observational study; OAD triple therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors; 2,4-thiazolidinedione; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Metformin/DPP4i/SGLT2i: Metformin + DPP4i 2-drug combination plus one of the SGLT-2i class of drugs.
  Interventions: Drug: SGLT2 inhibitor; Drug: DPP-4 inhibitor
- Metformin/DPP4i/TZD: Metformin + DPP4i 2-drug combination plus one of the TZD class of drugs.
  Interventions: Drug: Thiazolidinedione; Drug: DPP-4 inhibitor
- Metformin/SGLT2i/DPP4i: Metformin + SGLT2i 2-drug combination plus one of the DPP4i class of drugs.
  Interventions: Drug: SGLT2 inhibitor; Drug: DPP-4 inhibitor
- Metformin/SGLT2i/TZD: Metformin + SGLT2i 2-drug combination plus one of the TZD class of drugs.
  Interventions: Drug: SGLT2 inhibitor; Drug: Thiazolidinedione

INTERVENTIONS:
Drug: SGLT2 inhibitor — SGLT2 inhibitor class of drugs
  Groups: Metformin/DPP4i/SGLT2i; Metformin/SGLT2i/DPP4i; Metformin/SGLT2i/TZD
Drug: Thiazolidinedione — Thiazolidinedione class of drugs
  Groups: Metformin/DPP4i/TZD; Metformin/SGLT2i/TZD
Drug: DPP-4 inhibitor — DPP4 inhibitor class of drugs
  Groups: Metformin/DPP4i/SGLT2i; Metformin/DPP4i/TZD; Metformin/SGLT2i/DPP4i

SUMMARY:
A multicenter, prospective, non-interventional observation study to evaluate the safety and effectiveness of OAD triple therapy in Korean Type 2 diabetic mellitus patients.

DETAILED DESCRIPTION:
The study was designed as a multicenter, prospective, non-interventional, observational study in patients with type 2 diabetes mellitus who had inadequate glycemic control with conventional combination oral hypoglycemic agents including metformin.

Participants in this study will have type 2 diabetes mellitus with insufficient glycemic control on conventional combination therapy with a DPP-4i or SGLT2i oral hypoglycemic agent, including metformin, requiring the addition of one of the following: SGLT-2i, DPP-4i, or TZD.

The 3-drug combination therapy will be prescribed to subjects based on the medical judgment of the investigator based on the licensure of SGLT-2i, DPP-4i, or TZD(efficacy, dosing, precautions for use, etc.) in a real-world practice setting and all treatment and observation, including administration of medications and laboratory tests, will be based on the medical judgment of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes who are 19 years of age or older at the time of enrollment.
2. Continued DPP-4i or SGLT-2i oral hypoglycemic combination therapy with metformin for at least 8 weeks prior to enrollment.
3. 7.0% ≤ HbA1c < 10.0% based on laboratory tests performed within 4 weeks of enrollment.
4. Voluntarily give written informed consent after being told about the study.

Exclusion Criteria:

1. Patients with type 1 diabetes and secondary diabetes.
2. Patients receiving concomitant therapy with 3 or more oral hypoglycemic agents within 8 weeks of enrollment.
3. Requiring treatment with insulin, GLP-1, etc. in addition to oral hypoglycemic agents during the study.
4. End-stage renal disease and hemodialysis patients.
5. diabetic ketoacidosis Patients.
6. Pregnant and lactating women.
7. Patients who are contraindicated by any of the "Precautions for Use" in the license for the drug being administered during the study, given the observational nature of the study under routine practice.
8. Patients with a history of hypersensitivity to the investigational drug or any of its components or excipients.
9. Anyone else deemed by the investigator to be unsuitable for participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus whose glycemic control is inadequate on 2 oral hypoglycemic agents, including metformin.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Incidence of Adverse events in Triple Combination Therapy Including Metformin with SGLT-2i, DPP-4i, or TZD Class Drugs. | 24 month
  Safety assessment of triple combination therapy with Metformin SGLT2i or DPP4i and TZD class drugs(All adverse events occurring after the date of registration).

SECONDARY OUTCOMES:
Changes in HbA1c | 3, 6, (9), 12, 18, and 24 months
  Evaluation of HbA1c(%) Change Compared to Baseline in Each Combination Group
Changes in FPG | 3, 6, (9), 12, 18, and 24 months
  Evaluation of FPG(mg/dL) Change Compared to Baseline in Each Combination Group
Percentage of Subjects with HbA1c < 7.0% | 3, 6, (9), 12, 18, and 24 months
  Percentage of Subjects with HbA1c < 7.0% in Each Combination Group
Percentage of Subjects with HbA1c < 6.5% | 3, 6, (9), 12, 18, and 24 months
  Percentage of Subjects with HbA1c < 6.5% in Each Combination Group
Factors influencing HbA1c change at each endpoint for each combination group. | 24 month
  demographics, past hypoglycemic medications, hypoglycemic medication components and doses, duration of hypoglycemic medication, duration of disease, comorbidities, concomitant medications, etc.

OTHER OUTCOMES:
Changes in Weight | 3, 6, (9), 12, 18, 24 months
  Changes in Weight(kg) Compared to Baseline in Each Combination Group
Changes in waist circumference | 12 and 24 months
  Changes in waist circumference(cm) compared to Baseline in Each Combination Group (body composition in body water(L), protein(kg), minerals(kg), and body fat(kg))
Changes in Fatty Liver Index | 6, 12, 18, and 24 months
  Changes in Fatty Liver Index compared to Baseline in Each Combination Group
Changes in AST | 6, 12, 18, and 24 months
  Changes in AST(IU/L) Compared to Baseline in Each Combination Group
Changes in ALT | 6, 12, 18, and 24 months
  Changes in ALT(IU/L) Compared to Baseline in Each Combination Group
Changes Platelet Levels | 6, 12, 18, and 24 months
  Changes in Platelet(10^3/uL) Levels Compared to Baseline in Each Combination Group
Changes in Blood Lipid Levels(Total cholesterol, LDL-C, HDL-C, TG) | 6, 12, 18, and 24 months
  Change in Total cholesterol, LDL-C, HDL-C, TG(mg/dL) compared to Baseline in Each Combination Group
Changes in Insulin-Related Test Levels(HOMA-IR, HOMA-β) | 12 and 24 months
  Changes in HOMA-IR(%), HOMA-(%) compared to Baseline in Each Combination Group
Changes in eGFR | 12 and 24 months
  Changes in eGFR(mL/min/1.73m2) compared to Baseline in Each Combination Group
Changes in UACR | 12 and 24 months
  Changes in UACR(mg/g) compared to Baseline in Each Combination Group
Change in hsCRP | 12 and 24 months
  Change in hsCRP(mg/dL) compared to Baseline in Each Combination Group
Change in ProBNP(or NT-ProBNP) | 12 and 24 months
  Change in ProBNP(or NT-ProBNP)(pg/mL) compared to Baseline in Each Combination Group
Change in PP2 Compared to Baseline in Each Combination Group | 3, 6, (9), 12, 18, and 24 months
  Change in PP2(mg/dL) compared to Baseline in Each Combination Group.
Incidence Rate of Major Adverse Cardiovascular Events(MACE) | 24 month
  Incidence Rate of Major Adverse Cardiovascular Events(MACE) from Baseline to 24 Months for Each Combination Group
Incidence Rate of Diabetic Microvascular Events | 24 month
  Incidence Rate of Diabetic Microvascular Events from Baseline to 24 Months for Each Combination Group

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No